CLINICAL TRIAL: NCT00933101
Title: Prevalence of Oxidative Stress, Endothelial Dysfunction, Increased Carotid Artery Intima-media Thickness (cIMT) and Biomarkers of Vascular Inflammation in Adolescents With Type-1 Diabetes Mellitus (T1DM)
Brief Title: Vascular Inflammation in Adolescents With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Children's Mercy Hospital, Department of Endocrinology
Other Study IDs: 08 12-200E
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Type 1 Diabetes Mellitus; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HgbA1c <8: Adolescents with HgbA1c < or equal to 8% for the previous 12 months
- HgbA1c >10: Adolescents with HgbA1c > or equal to 10% for previous 12 months

SUMMARY:
The purpose of this study is to find out if diabetes damages the blood vessels of adolescents with good diabetes control compared to adolescents with less optimal control.

DETAILED DESCRIPTION:
Many published studies reveal that adult patients with T1DM can have early, silent and more advanced vessel wall thickness than normal subjects. This is influenced by the degree of their blood sugar control. If this is happening in adolescents, we want to know what proportion of adolescent children with type 1 diabetes show signs of early blood vessel damage. We also want to learn if these signs of damage are linked to other factors such as how long someone has had diabetes, blood sugar control or individual differences because of a difference in genetic make-up.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ages 12-18 years
* Tanner stage III-V
* T1DM > 2 years
* HgbA1c <8 or >10 for previous 2 years

Exclusion Criteria:

* Subjects with known history of hypercholesterolemia or family history of hypercholesterolemia
* Family history of premature cardiovascular disease
* Hypertension defined as subjects with blood pressure greater than the 90th percentile for age
* Anemia defined as Hgb <11.0 g/dl
* ADHD
* Congenital heart disease
* Pituitary tumor
* Known allergy to ultrasound gel
* Recent head injury
* Chromosomal abnormalities

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric Endocrinology clinic
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Determine the impact of glycemic control on vascular oxidative stress/inflammation in adolescents with Type 1 diabetes mellitus | 1 year

SECONDARY OUTCOMES:
To determine the impact of glycemic control and vascular oxidative stress/inflammation on vascular health in adolescents with T1DM | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ghufran Babar, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States